CLINICAL TRIAL: NCT02723318
Title: The Impact of Family Financial Support on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adam Schickedanz, Clinical Instructor in Pediatrics and Clinical Scholar, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLASchickedanzFCCog
Record Dates: First submitted 2016-03-25; First posted 2016-03-30 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Impaired Cognition
Keywords: Cognition; Financial Coaching; Social Determinants of Health; Socioeconomic Status
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financia Coaching & Social Services Referrals (Experimental): Enrollment in one-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Interventions: Behavioral: Financial Coaching; Behavioral: Access to Referrals to Social Services
- Social Services (Active Comparator): Enrollment in the control arm offers access to social services referrals.
  Interventions: Behavioral: Access to Referrals to Social Services

INTERVENTIONS:
Behavioral: Financial Coaching — One-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Arms: Financia Coaching & Social Services Referrals
Behavioral: Access to Referrals to Social Services

SUMMARY:
The investigators have partnered with financial coaching organizations to establish what the investigators have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on cognition using the Patient Reported Outcomes Measurement Information System (PROMIS) Cognition Short form 8a.

DETAILED DESCRIPTION:
Financial coaching is a new tool in the field of community development, but it has already demonstrated significant financial impact in a number of studies, including one randomized trial conducted by the Urban Institute. Financial coaching improves participant financial literacy, budgeting, saving for financial emergencies, and debt level. The investigators' project will help clinicians and the field of community economic development understand health and well-being through a new economic lens and assess the health-related impacts of the emerging field of financial coaching. The investigators have partnered with financial coaching organizations to establish what they have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on cognition using the Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Abilities Short Form.

Community-based participants will be recruited from South Los Angeles and randomized to receive either monthly financial coaching plus access to referral for social services (intervention) or access to referral for social services alone (control). Inclusion criteria include having dependents under age 18, having some form of income, and having a tax identification number (social security number or Individual tax identification number). Participants will be surveyed quarterly regarding their cognition using the PROMIS Cognitive Abilities Short Form 8-item survey.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they are caregivers/parents of one or more dependents, have some form of income, and have a tax identification number.

Exclusion Criteria:

* Inability to take part in financial coaching due to disability or primary language other than English or Spanish.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Cognition | Up to one year (if possible)
  Cognitive abilities will be assessed using the PROMIS Cognitive Abilities Survey short form 8a

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schickedanz, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- LIFT-LA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Participant consent did not include data sharing and there is no appropriate repository for data to be shared through.